CLINICAL TRIAL: NCT01443351
Title: Long-term Safety Study of Treatment With the Thrombopoietin Agonists Eltrombopag and Romiplostim in Patients With Primary Immune Thrombocytopenia (ITP)
Brief Title: Long-term Safety Study of Treatment With the Thrombopoietin Agonists Eltrombopag and Romiplostim in Patients With Immune Thrombocytopenia (ITP)
Status: Withdrawn | Type: Observational
Why Stopped: failure to recruit patients
Sponsor: Zealand University Hospital (Other)
Collaborators: Rigshospitalet, Denmark (Other); Odense University Hospital (Other)
Responsible Party: Principal Investigator, Sif Gudbrandsdottir, MD, Zealand University Hospital
Other Study IDs: TPO-SJ-227
Record Dates: First submitted 2011-09-13; First posted 2011-09-29 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Idiopathic Thrombocytopenic Purpura
Keywords: ITP; romiplostim; eltrombopag; bone marrow fibrosis; long-term safety
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic; Primary Myelofibrosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood samples will be collected, seru, plasma and mononuclear cells will be stored in a biobank for further research use
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- ITP patients: Patients with refractory ITP eligible for treatment with TPO-ra

SUMMARY:
Thrombopoietin Receptor Agonists (TPO-ra) are novel treatment modalities for patients with refractory Primary Immune Thrombocytopenia (ITP), but only few data are available for long-term effects of these drugs. In this observational study, effects and adverse effects including evaluation of bone marrow biopsies done at fixed intervals will be recorded from ITP patients treated with TPO-ra. For some patients, blood samples will be collected for research use.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with ITP
* platelet counts < 25 x10*9/L or < 50 x10*9/L with bleeding symptoms
* meets criteria for treatment with TPO-ra
* Females must use contraceptives when applicable for at least three months before inclusion

Exclusion Criteria:

* Pregnancy or nursing
* Former thromboembolic events excluding one incidence of deep venous thrombosis as complication to surgery or pregnancy or one incidence of cerebral embolism as complication to atrial fibrillation
* Liver insufficiency (for eltrombopag only)
* TPO-ra contraindications (e.g. allergy)
* TPO-ra treatments less than 6 months prior to inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patinets will be selected from Departments of Hematology
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Number of patients with sustained response at 6 months follow-up | 6 months
  Response is defined as platelet count > 30.000 mio/L and no bleeding

SECONDARY OUTCOMES:
Yearly response rates | 5 years
  Number of patients with response to treatment at 1, 2, 3, 4, and 5-year follow-up
Frequency of relapse | 5 years
Rate of splenectomy | 5 years
Development of reticulin fibrosis in bone marrow biopsies | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Hans Hasselbalch, Prof., MD, Principal Investigator — Department of Hematology, Copenhagen University Hospital Roskilde; Henrik Frederiksen, Dr., MD, Principal Investigator — Odense University Hospital; Sif Gudbrandsdottir, MD, Principal Investigator — Copenhagen University Hospital Roskilde
Locations (1):
- Copenhagen University Hospital Roskilde, Roskilde, Denmark